CLINICAL TRIAL: NCT04427137
Title: A Novel and Practical Accelerated Low-frequency Right-sided Stimulation Protocol as a Substitute for Patients With Bipolar Depression Needing Electroconvulsive Therapy During the COVID-19 Pandemic
Brief Title: Accelerated LFR for Bipolar Patients During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Daniel Blumberger, Medical Head and Co-Director, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 071-2020
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Bipolar Depression
Keywords: bipolar depression; transcranial magnetic stimulation; treatment resistance; low-frequency right-side stimulation
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerated LFR (Experimental): In the acute treatment phase, treatment will occur 8 times daily (50 min pause between treatments) on weekdays, until symptom remission is achieved (HRSD-24 score < to 10) or a maximum of 10 working days of daily treatment. In the tapering phase, treatments will be reduced to 2 treatment days per week for 2 weeks and then 1 treatment day per week for 2 weeks (4 weeks total). Patients that have responded to treatment will then enter the symptom-based relapse prevention phase including virtual check-in with study staff and a treatment schedule based on symptom level according to a modified relapse prevention algorithm that has been developed to prevent relapse after a successful course of ECT (known as the STABLE algorithm). The relapse prevention phase will last a maximum of 6 months.
  Interventions: Device: MagPro X100 Stimulator, B70 Fluid-Cooled Coil

INTERVENTIONS:
Device: MagPro X100 Stimulator, B70 Fluid-Cooled Coil — Treatment will occur 8 times per treatment day (50 min pause between treatments). Each treatment session will consist of a single LFR treatment, with 360 pulses of LFR delivered in one continuous train of 6 minutes at 1Hz at 120% of the patient's resting motor threshold.

SUMMARY:
The current study aims to assess the feasibility, acceptance and clinical outcomes of a practical high-dose LFR protocol, including tapering treatments and symptom-based relapse prevention treatments, in patients with bipolar depression previously responsive to ECT and patients needing urgent treatment due to symptom severity during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Treatment resistant bipolar depression is a leading cause of disability and socioeconomic burden of disease, and current treatment options all suffer from critical deficiencies of efficacy, capacity, or tolerability, especially given the current COVID-19 pandemic. rTMS and aLFR in particular has the potential to overcome many of these deficiencies, and is safe and well-tolerated. Taken together with the reported findings of other groups, aLFR may be feasible, tolerable, and capable of achieving comparable and potentially better remission rates than longer 20 to 30-day courses and it may also be beneficial to taper treatments and use symptom-based relapse prevention treatments in an aLFR protocol. Importantly, our pilot data in two patients previously responsive to ECT and data from the Cole et al. study suggest that accelerated rTMS may be a potential substitute for ECT as it may be possible to achieve remission in patients with severe depressive symptoms who would otherwise receive ECT. Furthermore, there is a burden of being able to provide care to as many people as possible based on severity of illness during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Currently are experiencing a bipolar depressive episode (bipolar disorder type 1 or 2) based on the MINI with or without psychotic symptoms
* Have previous response to ECT or high symptom severity warranting acute ECT in the opinion of one of the brain stimulation psychiatrists
* Are over the age of 18
* Pass the TMS adult safety screening (TASS) questionnaire
* Are voluntary and competent to consent to treatment

Exclusion Criteria:

* have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of substance dependence or abuse within the last 1 month
* Currently experiencing a mixed or manic episode (YMRS >12)
* have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
* have a lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder
* have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT or a febrile seizure of infancy or single seizure related to a known drug related event, cerebral aneurysm, significant head trauma with loss of consciousness for greater than 5 minutes
* have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
* currently take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy
* Lack of response to accelerated course of rTMS in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-01-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Proportion achieving remission on Hamilton Rating Scale for Depresion 24-it (HRSD-24) | Up to 10 days (From screening/baseline to end of the acute treatment)
  Less than or equal to 10
  This scale is used to quantify the severity of symptoms of depression Scale range: 0-76 (total score) Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)

SECONDARY OUTCOMES:
Change in Hamilton Rating Scale for Depresion 24-it (HRSD-24) | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
  This scale is used to quantify the severity of symptoms of depression Scale range: 0-76 (total score) Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Response on Hamilton Rating Scale for Depresion 24-it (HRSD-24) | Up to 10 days (From screening/baseline to end of the acute treatment)
  50% Reduction in score
  This scale is used to quantify the severity of symptoms of depression Scale range: 0-76 (total score) Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Change in Young Mania Rating Scale (YMRS) | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
  This scale is used to quantify the severity of symptoms of mania Scale range: 0-60 (total score) Lower scores indicate lower severity of manic symptoms (i.e., better outcome) Higher scores indicate higher severity of manic symptoms (i.e., worse outcome)
Remission on Patient Health Questionnaire (PHQ-9) | Up to 10 days (From screening/baseline to end of the acute treatment)
  Less than or equal to 4
  This scale is used to quantify the severity of symptoms of depression Scale range: 0-27 (total score) Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Response on Patient Health Questionnaire (PHQ-9) | Up to 10 days (From screening/baseline to end of the acute treatment)
  50% Reduction in score
  This scale is used to quantify the severity of symptoms of depression Scale range: 0-27 (total score) Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Change in Patient Health Questionnaire (PHQ-9) | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
  This scale is used to quantify the severity of symptoms of depression Scale range: 0-27 (total score) Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Remission on General Anxiety Disorder 7 item (GAD-7) | Up to 10 days (From screening/baseline to end of the acute treatment)
  Less than or equal to 4
  This scale is used to quantify the severity of symptoms of anxiety Scale range: 0-21 (total score) Lower scores indicate lower severity of anxiety symptoms (i.e., better outcome) Higher scores indicate higher severity of anxiety symptoms (i.e., worse outcome)
Response on General Anxiety Disorder 7 item (GAD-7) | Up to 10 days (From screening/baseline to end of the acute treatment)
  50% Reduction in score
  This scale is used to quantify the severity of symptoms of anxiety Scale range: 0-21 (total score) Lower scores indicate lower severity of anxiety symptoms (i.e., better outcome) Higher scores indicate higher severity of anxiety symptoms (i.e., worse outcome)
Change in General Anxiety Disorder 7 item (GAD-7) | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
  This scale is used to quantify the severity of symptoms of anxiety Scale range: 0-21 (total score) Lower scores indicate lower severity of anxiety symptoms (i.e., better outcome) Higher scores indicate higher severity of anxiety symptoms (i.e., worse outcome)
Remission on Beck Depression Inventory (BDI-II) | Up to 10 days (From screening/baseline to end of the acute treatment)
  Less than or equal to 12
  This scale is used to quantify the severity of symptoms of depression Scale range: 0-63 (total score) Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Response on Beck Depression Inventory (BDI-II) | Up to 10 days (From screening/baseline to end of the acute treatment)
  50% Reduction in Score
  This scale is used to quantify the severity of symptoms of depression Scale range: 0-63 (total score) Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Change on Beck Depression Inventory (BDI-II) | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
  This scale is used to quantify the severity of symptoms of depression Scale range: 0-63 (total score) Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
Remission on Beck Scale for Suicidal Ideation (SSI) | Up to 10 days (From screening/baseline to end of the acute treatment)
  Score of 0
  This scale is used to assess the presence or absence of suicidal ideation and the degree of severity of suicidal ideas Scale range: 0 - 38 (total score) Lower scores indicate lower severity of suicidal ideation (i.e., better outcome) Higher scores indicate higher severity of suicidal ideation (i.e., worse outcome)
Change on Beck Scale for Suicidal Ideation (SSI) | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
  This scale is used to assess the presence or absence of suicidal ideation and the degree of severity of suicidal ideas Scale range: 0 - 38 (total score) Lower scores indicate lower severity of suicidal ideation (i.e., better outcome) Higher scores indicate higher severity of suicidal ideation (i.e., worse outcome)
Change in WHO Disability Assessment Schedule (WHODAS) Range 0-38 | Up to 10 days (From screening/baseline to end of the acute treatment)
  changes in scores
Proportion of Patients Maintaining Response During Relapse Prevention | 24 weeks (Tapering and Relapse prevention phase)
  Includes number of treatment days needed and number going on to receive ECT

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blumberger, MD, Principal Investigator — CAMH
Locations (1):
- CAMH, Toronto, Ontario, Canada